CLINICAL TRIAL: NCT02322047
Title: Effect of Prazosin and Naltrexone on Personalized Script-Induced Alcohol Craving in Individuals With Alcohol Use Disorders With and Without Comorbid PTSD
Brief Title: Prazosin and Naltrexone (PaN) Study for Veterans With Alcohol Use Disorders
Acronym: PaN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: W81XWH-14-1-0025
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Results first posted 2020-12-29 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Alcohol Use Disorder; Posttraumatic Stress Disorder (PTSD)
Keywords: Alcohol Drinking; Craving; Drinking Behavior; Prazosin; Naltrexone; Adrenergic Alpha-1 Receptor Antagonists; Adrenergic Antagonists; Adrenergic Alpha-Antagonists; mu-Opioid Receptor Antagonist; Opioid Antagonist; Alcohol Use Disorder; Posttraumatic Stress Disorder; PTSD; Alcohol Treatment; Alcohol Dependence; Pharmacology Treatment; AUD; Alcohol Abuse; Substance Use Disorder; SUD; Substance Abuse; Addiction; Alcohol Addiction; Substance Addiction; Substance Dependence
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic; Alcohol Drinking; Drinking Behavior; Substance-Related Disorders; Behavior, Addictive | interventions — Prazosin; Naltrexone

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomized into one of four study conditions: Naltrexone/Prazosin (Nal/Praz), Naltrexone/Placebo (Nal/Pl), Prazosin/Placebo (Praz/Pl), and Placebo/Placebo (Pl/Pl). Randomization will be blocked by gender, PTSD status, and alcohol consumption goal (abstention vs. reduction) and will be conducted by a VA Puget Sound Research Pharmacist using randomization tables supplied by the study Principal Investigator (PI). The Research Pharmacist will have no additional contacts with the participants.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: No study staff, including the participants, will know which condition the participants are in. Only the Research Pharmacist will know the participants' conditions.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Praz/Nal (Experimental): Prazosin and Naltrexone.
  Prazosin will be taken following this titration schedule:
  Days 1-2: 1 mg @ 9PM Days 3-4: 1 mg @ 9AM, 3PM, 9PM Days 5-7: 2 mg @ 9AM, 3PM, 9PM Days 8-10: 2mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 11-14: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 15-42: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM
  Naltrexone will be taken from day 1 to day 42 at 9 PM. Dose: 50 mg.
  Interventions: Drug: Prazosin; Drug: Naltrexone
- Praz/Pl (Active Comparator): Prazosin and Placebo (Naltrexone)
  Prazosin will be taken following this titration schedule:
  Days 1-2: 1 mg @ 9PM Days 3-4: 1 mg @ 9AM, 3PM, 9PM Days 5-7: 2 mg @ 9AM, 3PM, 9PM Days 8-10: 2mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 11-14: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 15-42: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM
  Naltrexone Placebo will be taken from day 1 to day 42 at 9 PM. Dose: 50 mg.
  Interventions: Drug: Prazosin; Drug: Placebo (Naltrexone)
- Nal/Pl (Active Comparator): Naltrexone and Placebo (Prazosin)
  Prazosin Placebo will be taken following this titration schedule:
  Days 1-2: 1 mg @ 9PM Days 3-4: 1 mg @ 9AM, 3PM, 9PM Days 5-7: 2 mg @ 9AM, 3PM, 9PM Days 8-10: 2mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 11-14: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 15-42: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM
  Naltrexone will be taken from day 1 to day 42 at 9 PM. Dose: 50 mg.
  Interventions: Drug: Naltrexone; Drug: Placebo (Prazosin)
- Pl/Pl (Placebo Comparator): Placebo (Prazosin) and Placebo (Naltrexone)
  Prazosin Placebo will be taken following this titration schedule:
  Days 1-2: 1 mg @ 9PM Days 3-4: 1 mg @ 9AM, 3PM, 9PM Days 5-7: 2 mg @ 9AM, 3PM, 9PM Days 8-10: 2mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 11-14: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 15-42: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM
  Naltrexone Placebo will be taken from day 1 to day 42 at 9 PM. Dose: 50 mg.
  Interventions: Drug: Placebo (Prazosin); Drug: Placebo (Naltrexone)

INTERVENTIONS:
Drug: Prazosin — Prazosin Dosing Days 1-2: 1 mg @ 9PM Days 3-4: 1 mg @ 9AM, 3PM, 9PM Days 5-7: 2 mg @ 9AM, 3PM, 9PM Days 8-10: 2mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 11-14: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 15-42: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM
  Other Names: Minipress
  Arms: Praz/Nal; Praz/Pl
Drug: Naltrexone — Naltrexone Dosing Days 1-42: 50mg @ 9PM
  Arms: Nal/Pl; Praz/Nal
Drug: Placebo (Prazosin) — Placebo Dosing Days 1-2: 1 mg @ 9PM Days 3-4: 1 mg @ 9AM, 3PM, 9PM Days 5-7: 2 mg @ 9AM, 3PM, 9PM Days 8-10: 2mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 11-14: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 15-42: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM
  Other Names: Placebo
  Arms: Nal/Pl; Pl/Pl
Drug: Placebo (Naltrexone) — Placebo Dosing Days 1-42: 50mg @ 9PM
  Other Names: Placebo
  Arms: Pl/Pl; Praz/Pl

SUMMARY:
The purpose of this study is to evaluate whether the combination of prazosin and naltrexone will decrease alcohol cravings and drinking in individuals who have problems with alcohol and have used alcohol at risky levels compare to naltrexone and placebo (Nal/Pl), prazosin and placebo (Praz/Pl), and double-placebo (Pl/Pl). We hypothesize that those assigned to both prazosin and naltrexone would report significantly greater decreases in percent drinking days and heavy drinking days as well as significantly greater reduction in craving from pre to post-treatment than those assigned to either single medication or double-placebo.

Prazosin is a medication that is approved by the U.S. Food and Drug Administration (FDA) to treat people with high blood pressure. Some studies have shown that prazosin may also decrease nightmares and improve sleep in Veterans suffering from Posttraumatic Stress Disorder (PTSD). Animal studies have consistently found that prazosin is associated with decreased alcohol consumption and that the combination of prazosin and naltrexone outperforms either medication alone. The current study is evaluating an "off-label" use of prazosin to determine whether it is helpful in decreasing alcohol cravings and consumption among people with alcohol problems. "Off-label" means that the FDA has not approved the use of prazosin for alcohol problems.

Naltrexone is a medication that is FDA approved for treating alcohol problems.

This study is sponsored by the Department of Defense and the Congressionally Directed Medical Research Program (DoD/CDMRP). We expect approximately 120 participants in this study, which will run over approximately 4 years. Study participants will be involved in the study for 7 weeks, or until they complete the Final Assessment.

DETAILED DESCRIPTION:
In this double-blind, double-dummy, placebo-controlled study of prazosin and naltrexone, we will evaluate the combination of naltrexone and the noradrenergic medication prazosin (Nal/Praz) relative to naltrexone and placebo (Nal/Pl), prazosin and placebo (Praz/Pl), and double-placebo (Pl/Pl). Participants will undergo two craving inductions, one oriented towards relief craving and the other towards reward craving. Daily IVR (Interactive Voice Recording System) data on craving and consumption and PTSD symptomatology will be collected during the 7 days immediately following the initial assessment visit to establish a pre-medication baseline. One hundred twenty individuals with adequate IVR compliance and whose screening lab tests indicate it is safe for them to take the study medications will enter the medication phase of the study within 14 days of the initial assessment initiating prazosin/placebo as well as 50mg naltrexone/placebo treatment. Randomization will be blocked by gender, PTSD status, and desire to abstain vs. desire to cut down. Prazosin will be titrated to three times daily dosing (9 am: 4mg; 3pm: 4 mg; 9pm: 8mg) at the end of two weeks. Naltrexone will be taken once daily 50 mg/day with no titration schedule. The stable dose of both medications will continue for four more weeks and medication compliance will be evaluated through pill counts, the IVR daily monitoring, and riboflavin trace in urine analysis. On approximately day 42 participants will come into the lab for the craving inductions (there will be a two week window after day 42 in which participants may still be seen if scheduling issues arise). The order of the craving inductions will be counterbalanced, and their administration will be separated in time by 30 minutes to minimize carry over between them. Subjective responses to the craving inductions will be obtained via relief oriented craving items and reward oriented craving items from the Desire for Alcohol Questionnaire. Participants will then be assisted in returning their craving levels to baseline prior to debriefing. They will all be offered treatment referrals within the Veterans Affairs (VA) or in the community. Both prazosin and naltrexone can be safely discontinued without tapering.

ELIGIBILITY:
Inclusion Criteria:

1. Veteran of the U.S. military or National Guard Reserve.
2. Current AUD by DSM-5 criteria.
3. Heavy drinking (>14 drinks per week for females; > 21 drinks per week for males) for at least 2 weeks in the last 3 months and some drinking during the past two weeks OR binge drinking for at least 3 days in the last month (4+ drinks for females; 5+ drinks for males).
4. At least mild alcohol craving as assessed by the Pennsylvania Alcohol Craving Scale (PACS; score > 10) at baseline.
5. Age 18-80.
6. English fluency and literacy.
7. Trying or planning to try to cut down on or abstain from alcohol.
8. Good general medical health.
9. Capable of giving informed consent.

Exclusion Criteria:

1. Uncontrolled psychiatric disorder with psychotic symptoms or cognitive impairment.
2. If taking psychiatric medication, NOT on a stable dose for at least 30 days prior to randomization.
3. Any suicidal ideation in the past 7 days, plan or intent past 6 months, or any suicide attempt past year.
4. Homicidal ideation with plan and intent in the past 30 days.
5. Patient Health Questionnaire-9 (PHQ-9) endorsement of hopelessness or self-harm/SI and/or sum scale score ≥ 19.
6. Any use of prazosin or naltrexone past 30 days.
7. Currently taking disulfiram or acamprosate OR planning to take any of these medications (including prazosin or naltrexone) during the study.
8. Current moderate or severe substance use disorder (past 30 days) on any psychoactive substance other than alcohol, nicotine, or cannabis, OR use of any amphetamine or opioid-containing medications during the previous 30 days.
9. Significant acute or chronic medical illness
10. Preexisting hypotension (sys <100) or orthostatic hypotension (systolic drop of > 20 mmHg; after two minutes of standing, or any drop with dizziness).
11. Allergy or previous adverse reaction to naltrexone, prazosin, quinazolines, or other α-1 adrenergic blockers or use of other α -1 adrenergic blocker.
12. Women who are pregnant, breastfeeding, or of childbearing potential and not using a contraceptive method judged by the investigator to be effective.
13. Legal involvement that could interfere with study participation, including being court ordered for treatment.
14. Signs or symptoms of withdrawal at time of initial consent.
15. Any participation in an experimental drug study or any addiction study past 30 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-03-03 (Actual); Primary Completion 2018-10-10 (Actual); Study Completion 2018-10-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Simpson, Ph.D., Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Healthcare System, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berk E, Black J, Locastro J, Wickis J, Simpson T, Penk W. Traumatogenicity: effects of self-reported noncombat trauma on MMPIs of male Vietnam combat and noncombat veterans treated for substance abuse. J Clin Psychol. 1989 Sep;45(5):704-8. doi: 10.1002/1097-4679(198909)45:53.0.co;2-6. PMID 2808725
- [Background] Simpson TL, Westerberg VS, Little LM, Trujillo M. Screening for childhood physical and sexual abuse among outpatient substance abusers. J Subst Abuse Treat. 1994 Jul-Aug;11(4):347-58. doi: 10.1016/0740-5472(94)90045-0. PMID 7966505
- [Background] McCann BS, Simpson TL, Ries R, Roy-Byrne P. Reliability and validity of screening instruments for drug and alcohol abuse in adults seeking evaluation for attention-deficit/hyperactivity disorder. Am J Addict. 2000 Winter;9(1):1-9. doi: 10.1080/10550490050172173. PMID 10914288
- [Background] Simpson TL. Women's treatment utilization and its relationship to childhood sexual abuse history and lifetime PTSD. Subst Abus. 2002 Mar;23(1):17-30. doi: 10.1080/08897070209511472. PMID 12444358
- [Background] Simpson TL, Miller WR. Concomitance between childhood sexual and physical abuse and substance use problems. A review. Clin Psychol Rev. 2002 Feb;22(1):27-77. doi: 10.1016/s0272-7358(00)00088-x. PMID 11793578
- [Background] Simpson TL. Childhood sexual abuse, PTSD, and the functional roles of alcohol use among women drinkers. Subst Use Misuse. 2003 Jan;38(2):249-70. doi: 10.1081/ja-120017248. PMID 12625430
- [Background] Comtois KA, Tisdall WA, Holdcraft LC, Simpson T. Dual diagnosis: impact of family history. Am J Addict. 2005 May-Jun;14(3):291-9. doi: 10.1080/10550490590949479. PMID 16019979
- [Background] Simpson TL, Kivlahan DR, Bush KR, McFall ME. Telephone self-monitoring among alcohol use disorder patients in early recovery: a randomized study of feasibility and measurement reactivity. Drug Alcohol Depend. 2005 Aug 1;79(2):241-50. doi: 10.1016/j.drugalcdep.2005.02.001. Epub 2005 Feb 25. PMID 16002033
- [Background] Dobie DJ, Maynard C, Kivlahan DR, Johnson KM, Simpson T, David AC, Bradley K. Posttraumatic stress disorder screening status is associated with increased VA medical and surgical utilization in women. J Gen Intern Med. 2006 Mar;21 Suppl 3(Suppl 3):S58-64. doi: 10.1111/j.1525-1497.2006.00376.x. PMID 16637948
- [Background] Bowen S, Witkiewitz K, Dillworth TM, Chawla N, Simpson TL, Ostafin BD, Larimer ME, Blume AW, Parks GA, Marlatt GA. Mindfulness meditation and substance use in an incarcerated population. Psychol Addict Behav. 2006 Sep;20(3):343-7. doi: 10.1037/0893-164X.20.3.343. PMID 16938074
- [Background] Kaysen D, Simpson T, Dillworth T, Larimer ME, Gutner C, Resick PA. Alcohol problems and posttraumatic stress disorder in female crime victims. J Trauma Stress. 2006 Jun;19(3):399-403. doi: 10.1002/jts.20122. PMID 16788998
- [Background] Simpson T, Jakupcak M, Luterek JA. Fear and avoidance of internal experiences among patients with substance use disorders and PTSD: the centrality of anxiety sensitivity. J Trauma Stress. 2006 Aug;19(4):481-91. doi: 10.1002/jts.20128. PMID 16929503
- [Background] Simpson TL, Kaysen D, Bowen S, MacPherson LM, Chawla N, Blume A, Marlatt GA, Larimer M. PTSD symptoms, substance use, and vipassana meditation among incarcerated individuals. J Trauma Stress. 2007 Jun;20(3):239-49. doi: 10.1002/jts.20209. PMID 17597132
- [Background] Kaysen D, Dillworth TM, Simpson T, Waldrop A, Larimer ME, Resick PA. Domestic violence and alcohol use: trauma-related symptoms and motives for drinking. Addict Behav. 2007 Jun;32(6):1272-83. doi: 10.1016/j.addbeh.2006.09.007. Epub 2006 Nov 13. PMID 17098370

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was done from 03/03/2015 to 09/18/2018; however the last participant was recruited on 08/30/2018 because the rest of the interested individuals were not eligible. Participants were recruited primarily through letters that were sent to those whose medical records indicated they likely had an active Alcohol Use Disorder (AUD) and had not been prescribed the study medications. Other recruitment methods: flyers, VA TV monitors, and advertising in the local media.
Pre-assignment Details: Interested individuals called study staff and were screened for eligibility. Out of 200 phone screens, 97 individuals were eligible and invited to the screening visit. Of these, 21 did not show or were lost to follow up, 7 canceled their visit, and 8 declined the visit. Out of 61 individuals who came to screening, 31 were eligible and randomized.
Groups:
- Praz/Nal: Prazosin and Naltrexone.
  Prazosin will be taken following this titration schedule:
  Days 1-2: 1 mg @ 9PM Days 3-4: 1 mg @ 9AM, 3PM, 9PM Days 5-7: 2 mg @ 9AM, 3PM, 9PM Days 8-10: 2mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 11-14: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 15-42: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM
  Naltrexone will be taken from day 1 to day 42 at 9 PM. Dose: 50 mg.
  Prazosin: Prazosin Dosing Days 1-2: 1 mg @ 9PM Days 3-4: 1 mg @ 9AM, 3PM, 9PM Days 5-7: 2 mg @ 9AM, 3PM, 9PM Days 8-10: 2mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 11-14: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 15-42: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM
  Naltrexone: Naltrexone Dosing Days 1-42: 50mg @ 9PM
- Praz/Pl: Prazosin and Placebo (Naltrexone)
  Prazosin will be taken following this titration schedule:
  Days 1-2: 1 mg @ 9PM Days 3-4: 1 mg @ 9AM, 3PM, 9PM Days 5-7: 2 mg @ 9AM, 3PM, 9PM Days 8-10: 2mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 11-14: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 15-42: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM
  Naltrexone Placebo will be taken from day 1 to day 42 at 9 PM. Dose: 50 mg.
  Prazosin: Prazosin Dosing Days 1-2: 1 mg @ 9PM Days 3-4: 1 mg @ 9AM, 3PM, 9PM Days 5-7: 2 mg @ 9AM, 3PM, 9PM Days 8-10: 2mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 11-14: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 15-42: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM
  Placebo (Naltrexone): Placebo Dosing Days 1-42: 50mg @ 9PM
- Nal/Pl: Naltrexone and Placebo (Prazosin)
  Prazosin Placebo will be taken following this titration schedule:
  Days 1-2: 1 mg @ 9PM Days 3-4: 1 mg @ 9AM, 3PM, 9PM Days 5-7: 2 mg @ 9AM, 3PM, 9PM Days 8-10: 2mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 11-14: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 15-42: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM
  Naltrexone will be taken from day 1 to day 42 at 9 PM. Dose: 50 mg.
  Naltrexone: Naltrexone Dosing Days 1-42: 50mg @ 9PM
  Placebo (Prazosin): Placebo Dosing Days 1-2: 1 mg @ 9PM Days 3-4: 1 mg @ 9AM, 3PM, 9PM Days 5-7: 2 mg @ 9AM, 3PM, 9PM Days 8-10: 2mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 11-14: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 15-42: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM
- Pl/Pl: Placebo (Prazosin) and Placebo (Naltrexone)
  Prazosin Placebo will be taken following this titration schedule:
  Days 1-2: 1 mg @ 9PM Days 3-4: 1 mg @ 9AM, 3PM, 9PM Days 5-7: 2 mg @ 9AM, 3PM, 9PM Days 8-10: 2mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 11-14: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 15-42: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM
  Naltrexone Placebo will be taken from day 1 to day 42 at 9 PM. Dose: 50 mg.
  Placebo (Prazosin): Placebo Dosing Days 1-2: 1 mg @ 9PM Days 3-4: 1 mg @ 9AM, 3PM, 9PM Days 5-7: 2 mg @ 9AM, 3PM, 9PM Days 8-10: 2mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 11-14: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM Days 15-42: 4mg @ 9 AM, 3 PM; 8mg @ 9 PM
  Placebo (Naltrexone): Placebo Dosing Days 1-42: 50mg @ 9PM
Period: Overall Study
Arm/Group | Praz/Nal | Praz/Pl | Nal/Pl | Pl/Pl
Started | 8 | 7 | 7 | 9
Completed | 6 | 6 | 6 | 7
Not Completed | 2 | 1 | 1 | 2
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Only participants who completed the study or had an intention to treat (ITT) were included in analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Praz/Nal | Praz/Pl | Nal/Pl | Pl/Pl | Total
Number analyzed (Participants) | 7 | 7 | 7 | 8 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] — Age was collected in the screening visit using a demographic questionnaire.
  years | 51 (12.37) | 54.86 (9.08) | 54.43 (6.19) | 52.38 (10.72) | 53.14 (9.48)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender was collected in the screening visit using a demographic questionnaire.
  Participants
    Female | 1 | 0 | 0 | 1 | 2
    Male | 6 | 7 | 7 | 7 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity was collected in the screening visit using a demographic questionnaire.
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0 | 0
    Not Hispanic or Latino | 7 | 7 | 7 | 5 | 26
    Unknown or Not Reported | 0 | 0 | 0 | 3 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race was collected in the screening visit using a demographic questionnaire.
  Participants
    Asian/Pacific Islander | 1 | 0 | 0 | 0 | 1
    Black/African American | 0 | 1 | 2 | 2 | 5
    Native American/American Indian | 0 | 1 | 0 | 1 | 2
    White/Caucasian | 6 | 5 | 4 | 4 | 19
    Multiracial | 0 | 0 | 1 | 0 | 1
    Prefer not to answer | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 7 | 8 | 29
Percent drinking days (PDD) [Mean (Standard Deviation); unit: percentage of drinking days] — PDD was calculated based on self-reported drinking history collected via Form-90 in visit 2 (baseline visit). In this visit, participants reported their alcohol consumption from 90 days prior to their baseline visit until the day before their baseline visit. Drinking days were defined as days when participants consumed alcohol.
  percentage of drinking days | 73.10 (28.10) | 87.93 (19.87) | 64.44 (26.04) | 75.83 (21) | 75.34 (24.08)
Percent heavy drinking days (PHDD) [Mean (Standard Deviation); unit: percentage of heavy drinking days] — PHDD was calculated based on self-reported drinking history collected via Form-90 in visit 2 (baseline visit). In this visit, participants reported their alcohol consumption 90 days prior to their baseline visit until the day before their baseline visit if they drank 4 or more drinks (females) and 5 or more drinks (males).
  percentage of heavy drinking days | 54.99 (37.18) | 77.77 (28.63) | 47.62 (34.51) | 66.25 (33.60) | 61.81 (33.77)
Alcohol craving [Mean (Standard Deviation); unit: scores on scale] — Alcohol craving was assessed in the baseline and last visits using the Pennsylvania Alcohol Craving Scale (PACS). The PACS had 5 questions, where each question had six options presented in Likert Scales from 0 to 6, with 0 being the least and 6 being the highest possible option, thus the possible minimum and maximum values are 0 and 30, respectively. Higher scores mean higher craving.
  scores on scale | 18.50 (3.89) | 20.29 (6.68) | 16.71 (5.59) | 16.86 (5.76) | 18.10 (5.41)
Mean drinks per day of drinking [Mean (Standard Deviation); unit: drinks] — Average drinks per day of drinking were calculated based on self-reported drinking history collected via Form-90 in visit 2 (baseline visit). In this visit, participants reported their alcohol consumption from 90 days prior to their baseline visit until the day before their baseline visit. Drinking days were defined as days when participants consumed alcohol.
  drinks | 8.17 (5.40) | 11.88 (7.55) | 8.44 (3.97) | 13.88 (9.55) | 10.70 (7.12)

OUTCOME MEASURES:

1. Primary Outcome: Change in Percent Drinking Days (PDD) (Visit 8 PDD - Visit 2 PDD)
Description: PDD was calculated based on self-reported drinking history collected via Form-90. Drinking days were defined as days when participants consumed alcohol. Form-90 was completed by participants in visit 2 (baseline) and visit 8 (last visit). Form-90 collected in the baseline visit recorded participants' alcohol consumption from 90 days prior to their baseline visit until the day before their baseline visit. Form-90 collected in the last visit recorded participants' alcohol consumption from baseline until the day before their last visit. This outcome measures changes in PDD between visit 8 and visit 2. Per the protocol, visit 8 is scheduled to occur 42 days (± 7days) after visit 2. In reality, visit 8 occurred 35 to 76 days after visit 2 with the average of 45 days. The outliers were due to scheduling difficulties.
Time Frame: Visit 2 (baseline) and visit 8 (last visit). Per the protocol, visit 8 is scheduled to occur 42 days (± 7days) after visit 2. In reality, visit 8 occurred 35 to 76 days after visit 2 with the average of 45 days due to scheduling difficulties.
Population: Only participants who completed the study or had an intention to treat (ITT) were included in analyses.
Measure: Least Squares Mean (Standard Error); unit: percentage of drinking days
Arm/Group | Praz/Nal | Praz/Pl | Nal/Pl | Pl/Pl
Number analyzed (Participants) | 7 | 7 | 7 | 8
percentage of drinking days | -37 (10) | -9 (10) | -14 (10) | -15 (9)

2. Primary Outcome: Change in Percent Heavy Drinking Days (PHDD) (Visit 8 PHDD - Visit 2 PHDD)
Description: PHDD was calculated based on self-reported drinking history collected via Form-90. Heavy drinking days were defined as days when participants consumed 4 or more drinks for females and 5 or more drinks for males. Form-90 was completed by participants in the baseline and last visit. Form-90 collected in the baseline visit recorded participants' alcohol consumption 90 days prior to their baseline visit. Form-90 collected in the last visit recorded participants' alcohol consumption from baseline until the day before their last visit. This outcome measures changes in PHDD between visit 8 and visit 2. Per the protocol, visit 8 is scheduled to occur 42 days (± 7days) after visit 2. In reality, visit 8 occurred 35 to 76 days after visit 2 with the average of 45 days. The outliers were due to scheduling difficulties.
Time Frame: as for outcome 1
Population: Only participants who completed the study or had an intention to treat (ITT) were included in analyses.
Measure: Least Squares Mean (Standard Error); unit: percentage of heavy drinking days
Arm/Group | Praz/Nal | Praz/Pl | Nal/Pl | Pl/Pl
Number analyzed (Participants) | 7 | 7 | 7 | 8
percentage of heavy drinking days | -38 (17) | -8 (17) | -7 (17) | -13 (16)

3. Primary Outcome: Change in Alcohol Craving (Visit 8 PACS - Visit 2 PACS)
Description: Alcohol craving was assessed in visit 2 (baseline) and the last visit (visit 8) using the Pennsylvania Alcohol Craving Scale (PACS). The PACS had 5 questions, where each question had six options presented in Likert Scales from 0 to 6, with 0 being the least and 6 being the highest possible option, thus the possible minimum and maximum values are 0 and 30, respectively. Higher scores mean higher craving. This outcome measures the change in PACS scores between visits 2 and 8 (visit 8 PACS score - visit 2 PACS score). Per the protocol, visit 8 is scheduled to occur 42 days (± 7days) after visit 2. In reality, visit 8 occurred 35 to 76 days after visit 2 with the average of 45 days. The outliers were due to scheduling difficulties.
Time Frame: as for outcome 1
Population: Only participants who completed the study or had an intention to treat (ITT) were included in analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Praz/Nal | Praz/Pl | Nal/Pl | Pl/Pl
Number analyzed (Participants) | 7 | 7 | 7 | 8
score on a scale | -10.5 (2.4) | -4.6 (2.4) | -4.3 (2.4) | -3.5 (2.4)

4. Secondary Outcome: Change in Mean Drinks Per Day of Drinking (Visit 8 - Visit 2)
Description: Average drinks per day of drinking was calculated based on self-reported drinking history collected via Form-90. Drinking days were defined as days when participants consumed alcohol. Form-90 was completed by participants in visit 2 (baseline) and visit 8 (last visit). Form-90 collected in the baseline visit recorded participants' alcohol consumption 90 days prior to their baseline visit. Form-90 collected in the last visit recorded participants' alcohol consumption from baseline until the day before their last visit. This outcome reports the change in the mean drinks between visit 8 and visit 2. Per the protocol, visit 8 is scheduled to occur 42 days (± 7days) after visit 2. In reality, visit 8 occurred 35 to 76 days after visit 2 with the average of 45 days. The outliers were due to scheduling difficulties.
Time Frame: as for outcome 1
Population: Only participants who completed the study or had an intention to treat (ITT) were included in analyses.
Measure: Least Squares Mean (Standard Error); unit: drinks
Arm/Group | Praz/Nal | Praz/Pl | Nal/Pl | Pl/Pl
Number analyzed (Participants) | 7 | 7 | 7 | 8
drinks | -5.1 (1.7) | -2.2 (1.7) | -5.0 (1.7) | -3.7 (1.6)

ADVERSE EVENTS:
Time Frame: Participants went through 8 in-person visits (screening, baseline, and visits 3 to 8). Adverse events were collected after the baseline visit, the visit where participants were randomized and received medications, through 3 safety calls and 6 visits (visits 3 to 8). There was one safety call after the baseline visit, visit 3, and visit 4. Depending on whether a participant completed the study or not, adverse events were collected from 1 to 11 weeks.
Arm/Group | Praz/Nal | Praz/Pl | Nal/Pl | Pl/Pl
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7 | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7 | 0/7 | 0/9
Other Adverse Events (participants affected / at risk) | 5/8 | 3/7 | 3/7 | 3/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Praz/Nal (N=8) | Praz/Pl (N=7) | Nal/Pl (N=7) | Pl/Pl (N=9)
Dizziness (General disorders) | 4 | 0 | 1 | 2
Lightheadedness (General disorders) | 4 | 2 | 2 | 1
Drowsiness (General disorders) | 2 | 1 | 1 | 1
Lack of energy (General disorders) | 1 | 1 | 1 | 1
Weakness (General disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 1 | 1
Change in urination (Renal and urinary disorders) | 1 | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal symptoms (Gastrointestinal disorders) | 0 | 1 | 0 | 1 — Abdominal cramps, pain, and/or discomfort.
Decreased appetite (General disorders) | 0 | 0 | 0 | 2
Vivid dreams, nightmares (General disorders) | 0 | 0 | 1 | 0
Metallic taste in mouth (General disorders) | 0 | 1 | 0 | 0
Flushed (General disorders) | 0 | 1 | 0 | 0
Extreme energy, mania (General disorders) | 0 | 0 | 1 | 0
Insomnia, sleep disturbance (General disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-17): https://cdn.clinicaltrials.gov/large-docs/47/NCT02322047/Prot_SAP_000.pdf